CLINICAL TRIAL: NCT06298110
Title: The Effect of PRP on Wound Healing in High Risk Patients Undergoing Abdominal Hysterectomy
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Ahmed Mohammed El sayed, Doctor, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRP in Abdominal hysterectomy
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Wound Heal; Abdominal Wound; PRP
Keywords: PRP; Abdominal hysterectomy; Wound healing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): on the morning of surgery, 30 mL of venous blood will be drawn from the patient in anticoagulant-containing PRP tube for preparation of PRP solution. The drawn blood will be centrifuged at 1,200 rpm for 12 minutes to be separated into three layers: an upper layer that contains platelets and white blood cells, an intermediate thin layer (the buffy coat) that is rich in white blood cells, and a bottom layer that contains red blood cells. The upper and intermediate buffy layers will be transferred to an empty sterile tube. The plasma will be centrifuged again at 3,300 rpm for 7 minutes to help with the formation of soft pellets (erythrocytes and platelets) at the bottom of the tube. Pellets are homogenized in the lower third (5 mL) of the plasma to create the PRP. The prepared PRP solution will be transferred within sterile single use syringe (3cm) from the laboratory to the operation room, then applied and spread over the subcutaneous space before skin closure
  Interventions: Biological: Platelets Rich plasma of the same patient
- Control group (No Intervention): the patients received no topical treatment in the subcutaneous tissue or the skin before closure during surgery

INTERVENTIONS:
Biological: Platelets Rich plasma of the same patient — on the morning of surgery, 30 mL of venous blood will be drawn from the patient in anticoagulant-containing PRP tube for preparation of PRP solution. The drawn blood will be centrifuged at 1,200 rpm for 12 minutes to be separated into three layers: an upper layer that contains platelets and white blood cells, an intermediate thin layer (the buffy coat) that is rich in white blood cells, and a bottom layer that contains red blood cells. The upper and intermediate buffy layers will be transferred to an empty sterile tube. The plasma will be centrifuged again at 3,300 rpm for 7 minutes to help with the formation of soft pellets (erythrocytes and platelets) at the bottom of the tube. Pellets are homogenized in the lower third (5 mL) of the plasma to create the PRP. The prepared PRP solution will be transferred within sterile single use syringe (3cm) from the laboratory to the operation room, then applied and spread over the subcutaneous space before skin closure
  Arms: PRP group

SUMMARY:
To evaluate the effect of PRP on wound healing in high risk patients undergoing abdominal hysterectomy.

DETAILED DESCRIPTION:
Hysterectomy is one of the most common lines of surgical treatment of various uterine disorders as it provides definitive relief from the associated burdensome symptoms with an estimated prevalence of 13.1 per 10,000 women. The indications for hysterectomy include uterine leiomyomas (fibroid), dysfunctional uterine bleeding, endometrial adenomyosis, genital prolapse, massive postpartum hemorrhages and uterine cancers. Abdominal hysterectomy is still the most commonly used approach although there have been some preferences for vaginal and laparoscopic approaches.

Abdominal hysterectomy is associated with risk of complications. In high-risk women undergoing abdominal hysterectomy, wound healing can be particularly challenging due to a variety of factors, including poor tissue quality, compromised immune function, and underlying medical conditions.

Wound healing is a complex process that involves a series of events that are critical for the restoration of tissue integrity and function. Platelet-rich plasma (PRP) has emerged as a promising therapeutic option for enhancing wound healing in high risk patients. PRP is a concentrated source of platelets and growth factors derived from the patient's own blood. It has been shown to promote tissue regeneration and repair by stimulating cell proliferation, angiogenesis, and collagen synthesis. PRP has been used successfully in a variety of clinical settings, including orthopedics, dentistry, and dermatology.

PRP which contains concentrated growth factors have been reported to accelerate wound healing by30-40% giving a satisfactory outcome in the treatment of chronic skin and soft tissue lesions by supplying large amounts of growth factors and chemokines. When platelets become activated, they secrete Seven fundamental protein growth factors initiating all wound healing process, including platelet-derived growth factor (PDGF), epidermal growth factor (EGF), transforming growth factor (TGF), vascular endothelial growth factor (VEGF), Fibroblast growth factor (FGF), connective tissue growth factor (CTGF) & insulin like growth factor 1(ILGF 1), which participate in the acceleration of wound healing process.

A randomized controlled trial conducted by Tehranian et al. (2016) evaluated the use of PRP in high risk women after caesarian section. The study found that patients treated with PRP had significantly faster wound healing and a significant reduction in pain compared to those who received standard care. Similarly, another study by Fanning et al. (2007) investigated the use of PRP in women undergoing gynecologic surgery, there were no apparent adverse effects, and pain was significantly reduced.

In our study, we will investigate the effect of PRP on wound healing in high risk patients undergoing abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* - Female patients aged >18 years.
* Patients undergoing abdominal hysterectomy.
* Patients with a high risk of wound healing complications, including: obesity, diabetes mellitus, use of corticosteroid medication or smoking.

Exclusion Criteria:

* - Patients with hemoglobin (Hb) < 10 g/dL.
* Patients with platelet levels < 110 × 103/uL.
* Patients with coagulation disorders (on anticoagulant).
* Patients with malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2024-08-25 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
changes in wound healing | day 1, day 7, and day 30
  REEDA descriptive scale will assess degree of wound healing which formed of 4 points in a categorical score assessing 5 items of healing, redness, edema,ecchymosis, discharge approximation of the wound edges, each item is rated on a scale of 0-3 and total score may range between 0-15. lower scores indicating good healing

SECONDARY OUTCOMES:
Vancouver scar scale changes | day 1, day 7, and day 30
  Vancouver scar scale (VSS) use to detect changes of formation of keloids or hypertrophic scars. It assesses 4 subjective variables: vascularity, height/thickness, pliability, and pigmentation within a possible range of 0-14 for the total score. A lower score indicates better healing.
Visual Analog Scale changes | day 1, day 7, and day 30
  Pain was evaluated by the visual analog scale system (VAS) which assesses changes of pain via a continuous measurement instrument. The score is determined by measuring the distance (mm) between the no pain anchor to the point that the patient marks, providing a range of scores from 0-10. A higher score indicates greater pain intensity
Hospital readmission | 1 month post-operatively
  Need to hospital readmission due to wound complications
Infection | Up to 1 month
  Presence of infection after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa Bilal, Professor, Study Chair — Helwan University

REFERENCES:
- [Background] Akca A, Yilmaz G, Koroglu N. Platelet Indices as the Predictor of Antibiotics Response in Surgical Wound Infections Following Total Abdominal Hysterectomy. Sisli Etfal Hastan Tip Bul. 2019 Jun 24;53(2):132-136. doi: 10.14744/SEMB.2019.46693. eCollection 2019. PMID 32377071
- [Background] Fanning J, Murrain L, Flora R, Hutchings T, Johnson JM, Fenton BW. Phase I/II prospective trial of autologous platelet tissue graft in gynecologic surgery. J Minim Invasive Gynecol. 2007 Sep-Oct;14(5):633-7. doi: 10.1016/j.jmig.2007.05.014. PMID 17848327
- [Background] Gohar MM, Ali RF, Ismail KA, Ismail TA, Nosair NA. Assessment of the effect of platelet rich plasma on the healing of operated sacrococcygeal pilonidal sinus by lay-open technique: a randomized clinical trial. BMC Surg. 2020 Sep 22;20(1):212. doi: 10.1186/s12893-020-00865-x. PMID 32962673
- [Background] Madueke-Laveaux OS, Elsharoud A, Al-Hendy A. What We Know about the Long-Term Risks of Hysterectomy for Benign Indication-A Systematic Review. J Clin Med. 2021 Nov 16;10(22):5335. doi: 10.3390/jcm10225335. PMID 34830617
- [Background] Moscicka P, Przylipiak A. History of autologous platelet-rich plasma: A short review. J Cosmet Dermatol. 2021 Sep;20(9):2712-2714. doi: 10.1111/jocd.14326. Epub 2021 Jul 14. PMID 34214233
- [Background] Rodrigues M, Kosaric N, Bonham CA, Gurtner GC. Wound Healing: A Cellular Perspective. Physiol Rev. 2019 Jan 1;99(1):665-706. doi: 10.1152/physrev.00067.2017. PMID 30475656
- [Background] Tehranian A, Esfehani-Mehr B, Pirjani R, Rezaei N, Sadat Heidary S, Sepidarkish M. Application of Autologous Platelet-Rich Plasma (PRP) on Wound Healing After Caesarean Section in High-Risk Patients. Iran Red Crescent Med J. 2016 May 17;18(7):e34449. doi: 10.5812/ircmj.34449. eCollection 2016 Jul. PMID 27660723
- [Background] Veevers-Lowe J, Ball SG, Shuttleworth A, Kielty CM. Mesenchymal stem cell migration is regulated by fibronectin through alpha5beta1-integrin-mediated activation of PDGFR-beta and potentiation of growth factor signals. J Cell Sci. 2011 Apr 15;124(Pt 8):1288-300. doi: 10.1242/jcs.076935. Epub 2011 Mar 23. PMID 21429937
- See also: Impact of hysterectomy on uterine cancer incidence rates in Egypt — https://doi.org/10.15406/ogij.2021.12.00547